CLINICAL TRIAL: NCT05015959
Title: Analysis of Surgical Mortalities Using the Fishbone Model for Quality Improvement
Status: Completed | Type: Observational
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Maeyane Stephens Moeng, Prof, University of Witwatersrand, South Africa
Other Study IDs: M190122
Record Dates: First submitted 2021-08-03; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Complication of Surgical and Medical Care, Unspecified
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mortality outcomes: mortality classification into preventable, potentially preventable and non-prevenatable
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — quality
  Other Names: mortality outcomes

SUMMARY:
Retrospective data analysis of mortalities and the evaluation of the quality of care offered, using the Fishbone method.

DETAILED DESCRIPTION:
Evaluation of mortalities seen between 01 January 2017 and 31 December 2018. Analysis of the mortality decision into preventable, non-preventable and potentially preventable categories. Identifying the associated risk factors and co-morbidities in a single centre study in Johannesburg. Further analysing was performed on the subset of preventable mortalities and further do the fishbone model of quality of care. RedCap data was utilized for all data points. A further comparison was done to the MNM classification based on the team and an independent senior surgeon.

ELIGIBILITY:
Inclusion Criteria: All mortality of patients seen in the Department who were 18yrs or older

-

Exclusion Criteria:

* incomplete data death in the Emergency department

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all adults 18 years or older that presented to our institution and died withing the study period.
Sampling Method: Non-Probability Sample
Enrollment: 859 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
mortality outcomes | study period (Jan 2017 to Dec 2018)
  in-hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Maeyane Moeng, MBBCH, FCS, Principal Investigator — University of Witwatersrand, South Africa
Locations (1):
- Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Undecided